CLINICAL TRIAL: NCT00086060
Title: Locus of Pain Control: Neural Substrates and Modifiability
Brief Title: Pain Management Techniques for Fibromyalgia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, David A. Williams, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAMS-121; R01AR050044-01A1 (NIH)
Record Dates: First submitted 2004-06-22; First posted 2004-06-23 (Estimated); Last update posted 2011-10-10 (Estimated); Status verified 2011-10

CONDITIONS: Fibromyalgia
Keywords: Internal-External Control; Magnetic Resonance Imaging; fMRI; Exercise; Relaxation
MeSH Terms: conditions — Fibromyalgia; Motor Activity | interventions — Relaxation Therapy; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 - Relaxation Training (Experimental): Participants will receive relaxation training and standard care for FM
  Interventions: Behavioral: Relaxation training
- 2 Exercise Regimen (Experimental): Participants will receive an exercise regimen and standard care for FM
  Interventions: Behavioral: Exercise regimen
- 3 Standard Care (Active Comparator): Participants will receive standard of care for FM
  Interventions: Behavioral: Standard Care
- 4 Health Controls (No Intervention): Health participants will act as a control

INTERVENTIONS:
Behavioral: Exercise regimen — Aerobic Exercise is a self-management technique that increases personal control over pain by enhancing physical fitness. Patients will be encouraged to choose activities best suited to their tastes and current lifestyle, incorporating lifestyle physical activities (climbing stairs, household chores, etc) and more traditional exercise activities (walking, cycling, etc.). Subjects will use ratings of perceived exertion (RPE) to guide their effort. The intervention will consist of two-hours of face-to-face contact followed by weekly telephone contact for 8 weeks. Face-to-face contract will include receiving a standardized instruction manual for exercise, a demonstration on how to perform relaxation, and tailoring homework assignments to be monitored on the weekly phone call.
  Arms: 2 Exercise Regimen
Behavioral: Relaxation training — Relaxation is a self-management technique that increases personal control over pain by relaxing tense muscles, allowing the body to rest, and improving mental clarity through concentration and attention and has a great deal of empirical research supporting its effectiveness as a means of pain management. A variety of relaxation skills will be taught with some being based on muscle relaxation, and others focused more on cognitive relaxation and imagery. The intervention will consist of two-hours of face-to-face contact followed by weekly telephone contact for 8 weeks. Face-to-face contract will include receiving a standardized instruction manual for relaxation, a demonstration on how to perform relaxation, and tailoring homework assignments to be monitored on the weekly phone call.
  Arms: 1 - Relaxation Training
Behavioral: Standard Care — Participants in the standard care control group will not receive any additional intervention beyond that which they are receiving from their routine health care professional.
  Arms: 3 Standard Care

SUMMARY:
Pain management techniques may influence how the brain processes pain and may help patients with fibromyalgia (FM), a chronic pain condition. This study will train patients with FM to use pain management techniques. Investigators will use brain scanning (functional magnetic resonance imaging, or fMRI) technology to identify changes in how a patient's brain processes pain over time. This study is primarily interested in examining cortical response to different behavioral interventions.

DETAILED DESCRIPTION:
FM is a chronic pain condition that has no cure, and drugs are only partially successful in managing its symptoms. Many people with FM utilize nondrug management methods, such as exercise, for symptom relief. Nondrug methods can be quite effective, but some patients find it difficult to use these methods consistently. This study will determine which nondrug methods relieve FM symptoms by examining patients' brains after exercise or relaxation techniques. Preliminary data indicate that beliefs about one's personal ability to control pain result in use of differential neural mechanisms to process pain. This study will use fMRI, a tool for visualizing pain-processing patterns, to gain insights into how exercise and relaxation techniques modify pain processing in patients with FM.

There are four arms in this study. All participants with FM will be randomly assigned to one of three study arms. Participants in Arm 1 will receive relaxation training to supplement standard care for FM. Arm 2 participants will be prescribed an exercise regimen to supplement standard care. Participants in Arm 3 will receive standard care only. Arm 4 is a healthy control group, which will be followed during the 8-week intervention period.

At baseline, all participants will undergo blood collection and physical examination and will complete questionnaires about demographics, treatment history, symptoms, functional status, affective status, and beliefs about pain. They will also undergo a baseline fMRI imaging study, combined with evoked pressure pain testing, to evaluate differences in neural mechanisms involved in pain processing. Patients in Arms 1 and 2 will then attend one face-to-face training session with a therapist, followed by phone contact over the next 8 weeks. Participants will be asked to record pain and adherence to treatment on an electronic diary. After 8 weeks, all study participants will undergo a second fMRI scan, blood collection, and physical examination, and will complete questionnaires similar to those completed at baseline.

ELIGIBILITY:
Note: Given that this study requires participation in a number of appointments and reimbursement will not be made for travel expenses, individuals residing more than 100 miles from Ann Arbor are not encouraged to participate in this project.

Inclusion Criteria for Arms 1, 2, and 3:

* Diagnosis of fibromyalgia based on the criteria outlined by the American College of Rheumatology
* Standard medical care for fibromyalgia with the referring physician for at least the past 3 months

Exclusion Criteria for All Participants:

* Severe physical impairment that would prevent the participant from receiving either of the nondrug interventions (e.g., complete blindness, deafness, paraplegia) or coexisting physical impairments that could be harmed by light exercise (e.g., sprained ankle, neck injury)
* Morbid obesity
* Autoimmune disease
* Cardiopulmonary disorders (e.g., angina, congestive heart failure, COPD, chronic asthma)
* Uncontrolled endocrine or allergic disorders (e.g., thyroid dysfunction, Type I diabetes)
* Cancer within the past 2 years
* Current psychiatric disorder involving a history of psychosis (e.g., schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder), current suicide risk or suicide attempt within 2 years of study entry, or substance abuse within 2 years of study entry. Participants with mood disorders will not be excluded.
* Any pending or active disability associated with fibromyalgia (e.g., SSI, Workers' Compensation)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2004-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Change in clinical pain | Measured at Week 8
Change in activation pattern in fMRI | Measured at Week 8
Change in locus of control | Measured at Week 8

SECONDARY OUTCOMES:
Improvement in symptoms | Measured at Week 8
Improvement in function | Measured at Week 8
Improvement in mood | Measured at Week 8

CONTACTS AND LOCATIONS:
Overall Officials: David A. Williams, PhD, Principal Investigator — Chronic Pain and Fatigue Research Center, University of Michigan
Locations (1):
- Chronic Pain and Fatigue Research Center, University of Michigan, Ann Arbor, Michigan, United States